CLINICAL TRIAL: NCT00701051
Title: Aging, Angiogenesis and Metabolic Responses to Aerobic Exercise
Brief Title: Exercise Training and Glucose Metabolism in Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: University of Maryland (Other); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDA-2-039-08S; H-27940 (Other: IRB); 5P30AG028747-05 (NIH)
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2015-04-06 (Estimated); Last update posted 2015-04-06 (Estimated); Status verified 2015-03

CONDITIONS: Type 2 Diabetes Mellitus; Impaired Glucose Tolerance (Prediabetes)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Older adults, normal glucose tolerance
  Interventions: Behavioral: Aerobic exercise training; Behavioral: Detraining (cessation of exercise)
- Arm 2 (Experimental): Older adults, impaired glucose tolerance
  Interventions: Behavioral: Aerobic exercise training; Behavioral: Detraining (cessation of exercise)

INTERVENTIONS:
Behavioral: Aerobic exercise training — 24 weeks of aerobic exercise training: 3 times per week, 60 minutes per session, at 70% of maximal aerobic capacity
Behavioral: Detraining (cessation of exercise) — Cessation of exercise for 2 weeks

SUMMARY:
Diabetes and its associated complications affect more than 20 million Americans, and the prevalence of type 2 diabetes and impaired glucose tolerance rises dramatically with age such that 40% of Americans over age 60 are affected. In older adults, glucose metabolism may be affected by reduced skeletal muscle capillary supply, which limits insulin, glucose, and oxygen delivery to skeletal muscle. Reduced capillary supply to skeletal muscle is found in older individuals with impaired glucose tolerance and we hypothesize that this is due to reduced vascular growth factor expression, and chronic inflammation. Further, we hypothesize that reversal of a sedentary lifestyle through aerobic exercise training will increase insulin signaling and vascular growth factor expression, as well as decrease inflammation, to increase capillary supply to skeletal muscle, which contributes to improved glucose metabolism in older adults. This study will: 1) Determine the mechanisms underlying reduced skeletal muscle capillarization in older adults with impaired glucose tolerance; and 2) Determine the effect of aerobic exercise training-induced increases in skeletal muscle capillarization on glucose metabolism in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years
* Non-smoker >2 years
* Body mass index = 18-35 kg/m2

Exclusion Criteria:

* History of CAD or cerebrovascular disease that would preclude exercise
* Implantable defibrillator
* Active cancer
* Chronic pulmonary, thyroid, renal, liver, or hematological disease
* HIV positive or prone to malnutrition
* Sickle cell anemia
* Type 1 diabetes, or currently on medication to treat type 2 diabetes
* Poorly-controlled type 2 diabetes
* Poorly-controlled hypertension
* Taking medications including: beta-blockers, oral steroids, warfarin, certain statins, hormone replacement therapy (HRT), oral contraceptives (OCP), thiazolidinediones (TZD), or chronic steroids or nonsteroidal analgesics (NSAIDS) that may not be safely discontinued temporarily for specific procedures (i.e. for 72 hours prior)
* Allergic to lidocaine or heparin
* Recent weight change (>5kg in 3 months)
* Currently pregnant or nursing
* Physical impairment limiting exercise
* Dementia or unstable clinical depression

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-10; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J. Prior, PhD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (1):
- VA Maryland Health Care System, Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Prior SJ, Goldberg AP, Ortmeyer HK, Chin ER, Chen D, Blumenthal JB, Ryan AS. Increased Skeletal Muscle Capillarization Independently Enhances Insulin Sensitivity in Older Adults After Exercise Training and Detraining. Diabetes. 2015 Oct;64(10):3386-95. doi: 10.2337/db14-1771. Epub 2015 Jun 11. PMID 26068543

RESULTS

PARTICIPANT FLOW:
Groups:
- Older Adults - Normal Glucose Tolerance: Normal Glucose Tolerance. Participants assigned to group after Period 1: Screening
- Older Adults - Impaired Glucose Tolerance: Impaired Glucose Tolerance. Participants assigned to group after Period 1: Screening
Period: Screening
Arm/Group | Older Adults | Older Adults - Normal Glucose Tolerance | Older Adults - Impaired Glucose Tolerance
Started | 90 (Arm assignment not known until baseline testing; both arms included in this number) | 0 | 0
Completed | 31 (Arm assignment not known until baseline testing; both arms included in this number) | 0 | 0
Not Completed | 59 | 0 | 0
Not completed — Failed Screening | 40 | 0 | 0
Not completed — Time conflicts | 19 | 0 | 0
Period: Exercise Intervention
Arm/Group | Older Adults | Older Adults - Normal Glucose Tolerance | Older Adults - Impaired Glucose Tolerance
Started | 0 (Participants assigned to Normal or Impaired glucose tolerance arm after screening.) | 19 (Participants assigned to group after Period 1: Screening) | 12 (Participants assigned to group after Period 1: Screening)
Completed | 0 | 14 | 9
Not Completed | 0 | 5 | 3
Not completed — time conflict; non-study related illness | 0 | 5 | 3
Period: Detraining Intervention (Optional)
Arm/Group | Older Adults | Older Adults - Normal Glucose Tolerance | Older Adults - Impaired Glucose Tolerance
Started | 0 | 6 (Participation in this period was optional.) | 6 (Participation in this period was optional.)
Completed | 0 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Older Adults - Normal Glucose Tolerance: Normal Glucose Tolerance
- Older Adults - Impaired Glucose Tolerance: Impaired Glucose Tolerance
- Total: Total of all reporting groups
Arm/Group | Older Adults - Normal Glucose Tolerance | Older Adults - Impaired Glucose Tolerance | Total
Number analyzed (Participants) | 19 | 12 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (7) | 60 (8) | 60 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 10 | 6 | 16

OUTCOME MEASURES:

1. Primary Outcome: Baseline Glucose Utilization
Description: Insulin-stimulated glucose uptake
Time Frame: baseline
Measure: Mean (Standard Error); unit: µmol/kgFFM/pmol insulin/min
Arm/Group | Older Adults - Normal Glucose Tolerance | Older Adults - Impaired Glucose Tolerance
Number analyzed (Participants) | 19 | 12
µmol/kgFFM/pmol insulin/min | 0.0062 (.00008) | 0.0035 (0.0004)

2. Secondary Outcome: Baseline 2-hour Postprandial Glucose
Time Frame: baseline
Measure: Mean (Standard Error); unit: mg/dl
Arm/Group | Older Adults - Normal Glucose Tolerance | Older Adults - Impaired Glucose Tolerance
Number analyzed (Participants) | 19 | 12
mg/dl | 107 (2) | 160 (10)

3. Primary Outcome: Glucose Utilization (Pre/Post Intervention)
Description: Insulin-stimulated glucose uptake
Time Frame: baseline, 24 weeks, 26 weeks
Population: Glucose tolerance data were analyzed as a continuous variable (combining Arms) as opposed to categorical (i.e., within each Arm) due to the sample size of this pilot study; thus, data are reported for the entire group of participants.
Measure: Mean (Standard Error); unit: µmol/kgFFM/pmol insulin/min
Groups:
- Older Adults: Normal and Impaired Glucose Tolerance
Arm/Group | Older Adults
Number analyzed (Participants) | 12
µmol/kgFFM/pmol insulin/min
  Baseline | 0.041 (0.005)
  24-week | 0.052 (0.006)
  26-week | 0.048 (0.005)

4. Secondary Outcome: 2-hr Post-prandial Plasma Glucose Level
Time Frame: baseline, 24 weeks, 26 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Older Adults
Number analyzed (Participants) | 12
mg/dL
  Baseline | 173 (8)
  24-week | 153 (16)
  26-week | 142 (19)

5. Secondary Outcome: Baseline Cardiorespiratory Fitness
Description: maximal oxygen consumption
Time Frame: baseline
Measure: Mean (Standard Error); unit: L/min
Arm/Group | Older Adults - Normal Glucose Tolerance | Older Adults - Impaired Glucose Tolerance
Number analyzed (Participants) | 19 | 12
L/min | 2.2 (0.3) | 1.7 (0.2)

6. Primary Outcome: Baseline Skeletal Muscle Capillarization
Time Frame: baseline
Measure: Mean (Standard Error); unit: capillaries/mm2
Arm/Group | Older Adults - Normal Glucose Tolerance | Older Adults - Impaired Glucose Tolerance
Number analyzed (Participants) | 19 | 12
capillaries/mm2 | 313 (13) | 246 (8)

7. Primary Outcome: Skeletal Muscle Capillarization (Pre/Post Intervention)
Time Frame: baseline, 24 weeks, 26 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: capillaries/mm2
Arm/Group | Older Adults
Number analyzed (Participants) | 12
capillaries/mm2
  Baseline | 289 (12)
  24-week | 341 (21)
  26-week | 361 (10)

8. Secondary Outcome: Cardiorespiratory Fitness
Description: Maximal oxygen consumption
Time Frame: baseline, 24 weeks, 26 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: L/Min
Arm/Group | Older Adults
Number analyzed (Participants) | 12
L/Min
  Baseline | 1.8 (0.1)
  24-week | 2.3 (0.5)
  26-week | 2.2 (0.5)

9. Secondary Outcome: Body Composition (%Fat)
Time Frame: baseline, 24 weeks
Population: as for outcome 3
Measure: Mean (Standard Error); unit: percentage of fat
Arm/Group | Older Adults
Number analyzed (Participants) | 12
percentage of fat
  Baseline | 35 (3)
  24-week | 33 (3)

ADVERSE EVENTS:
Groups:
- Older Adults: Glucose tolerance data were analyzed as a continuous variable (combining Arms) as opposed to categorical (i.e., within each Arm); thus, data are reported for the entire group of participants.
Arm/Group | Older Adults
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 1/90
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Older Adults (N=90)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) — Fall due to distraction while walking

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes